CLINICAL TRIAL: NCT04126772
Title: Multimodal Imaging of MS Reveals the Smoldering Inflammation
Acronym: PLAQ-MS
Status: Active, not recruiting | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: PLAQ-MS
Record Dates: First submitted 2019-08-05; First posted 2019-10-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and faecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Active MS patients: 10 MS patients with an active lesion of 0,5 cm diameter
- Healthy controls: 20 healthy controls
- SPMS patients: 10 SPMS patients

SUMMARY:
To evaluate active MS plaque evolution with conventional MRI, QSM-post processing, TSPO-PET imaging and P2X7-PET imaging.

DETAILED DESCRIPTION:
Objective: To establish the QSM-MRI-method as a part of MS-patient research protocol in TPC and to quantify the time and space dependent correlation of QSM-MRI signal and PET-imaging signal with both 11C-PK11195 and 11C-SMW139 radioligands in the brain of MS-patients with active disease, secondary progressive MS-patients and healthy controls.

Background: In MS brain the inflammatory lesions change over time from active to chronic active and finally to chronic inactive plaques. Conventional MRI-imaging is used to detect the lesions but it is not able to differentiate the plaque types. The most acute lesions with blood-brain-barrier defect can be identified using conventional MRI and gadolinium enhancing, but follow-up of the later plaque development with microglial activation at plaque edge is not possible using MRI. Furthermore, the diffuse microglial activation in the NAWM is not detectable with conventional MRI.

In previous studies it has been shown that chronic active plaques have a rim of active microglial cells around them. With QSM-MRI method it is possible to detect and quantify these iron containing active microglia cells around the chronic active plaque. Active microglial cells can also be detected with PET imaging and TSPO-binding radioligand 11C-PK11195 or P2X7 binding radioligand 11C-SMW139. The investigators expect that the microglial activation signals detected with QSM-MRI and PET are co-localized and that these methods would help to differentiate the plaque types and to evaluate the MS plaque evolution.

Study population: 10 MS-patients with acute gadolinium enhancing ≥0,5cm diameter lesion will be imaged at baseline and 4 and 18 months after that. For comparison 10 secondary progressive patients and 20 healthy controls will be imaged at baseline.

Methods: Clinical evaluation, brain QSM-MRI and PET imaging with 11C-PK11195 radiotracer will be performed at baseline, 4 months and 18 months. PET imaging with 11C-CSMW139 radiotracer will be performed at 4 months and 18 months.

For healthy controls, brain QSM-MRI, PET imaging with 11C-PK11195 radiotracer and PET imaging with 11C-SMW139 radiotracer will be performed at baseline. For 12 healthy controls a test-retest imaging with 11C-SMW139 radiotracer will be performed.

ELIGIBILITY:
Inclusion Criteria

Active MS-patients:

* Informed consent form
* At least one 0,5 cm diameter active gadolinium enhancing lesion detected lately
* Diagnosed MS-disease according to McDonald criteria

SPMS patients

* Informed consent form
* Diagnosed MS-disease according to McDonald criteria
* SPMS disease

Healthy controls:

* Informed consent form
* healthy
* age and sex matched with MS-patients in RRMS and SPMS groups

Exclusion Criteria

MS-patients:

* Patients suffering from another brain disease or other autoimmune disease in addition to multiple sclerosis
* Steroid treatment 4 weeks prior to the scan
* Significant pathology in the MRI scan other than MS-related lesions
* Patients suffering from claustrophobia or panic disorder, or patients who have exhibited hypersensitivity of PET markers (practical obstacle to the scan)
* Exposure to experimental radioactivity in the last 12 months such that the dosimetry threshold would be exceeded due to participation in the study
* Age over 70

Healthy controls:

* autoimmune disease, CNS disease or other serious disease
* Steroid treatment 4 weeks prior to the scan or other regular medication
* persons suffering from claustrophobia or panic disorder, or persons who have exhibited hypersensitivity of PET markers (practical obstacle to the scan)
* Exposure to experimental radioactivity in the last 12 months such that the dosimetry threshold would be exceeded due to participation in the study
* Age over 70

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will recruit MS patients with active disease and at least 0,5 cm diameter gadolinium enhancing lesion who are followed-up at the Neurology Outpatient Clinic at the Turku University Hospital. The study will not interfere with the initiation or dosage of medication in any manner. For comparison the study will also recruit healthy subjects and secondary progressive MS-patients.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-02-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
11C-PK11195 binding in MS patient brain | Baseline, 4 months 18 months
  Change in microglia-activity in MS patients during 18 months as measured by [11C]PK11195 PET imaging
11C-SMW139 binding in MS patient brain | Baseline, 4 months 18 months
  Change in microglia-activity in MS patients during 18 months as measured by [11C]SMW139 PET imaging
QSM-signal in MS patient brain | Baseline, 4 months 18 months
  Change in microglia-activity in MS patients during 18 months as measured by QSM-MRI

SECONDARY OUTCOMES:
11C-PK11195 binding in healthy control brain | Baseline
  Change in microglia-activity in healthy controls during 18 months as measured by PET imaging and [11C]PK11195
11C-SMW139 binding in healthy control brain | Baseline
  Change in microglia-activity in healthy controls during 18 months as measured by PET imaging [11C]SMW139
QSM-signal in healthy control brain | Baseline
  Change in microglia-activity in healthy controls during 18 months as measured by QSM-MRI
MRI metrics | Baseline, 4 months, 18 months
  To evaluate lesion load of the white matter MS plaques
EDSS | Baseline, 4 months, 18 months
  Expanded Disability Status Scale. The scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability.
MSFC | Baseline, 4 months, 18 months
  Multiple Sclerosis Composite Score which consists of three assessments of walking speed, processing speed and finger dexterity. The scores are combined to provide a Z-score. Lower scores represent greater abnormality.
Fatigue severity scale | Baseline, 4 months, 18 months
  Fatigue Severity Scale is a self-reported, 9-item fatigue scale. Participants rate all 9 items on a 7-point Likert scale (1-2-3-4-5-6-7) depending on how appropriate they felt the statement applied to them over the preceding week. The total score is calculated by adding up the answer from each item and divide by 9. Lower scores indicate better outcomes. Maximum score is 7.
Modified Fatigue Impact Scale | Baseline, 4 months, 18 months
  The Modified Fatigue Impact Scale is a self-report survey that contains 21 items. Each item is rated 0-4. Higher scores indicate a greater impact of fatigue on a person's activities.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Airas, MD,professor, Principal Investigator — Turku University Hospital, division of clinical neurosciences
Locations (1):
- Turku PET Centre, Turku, Southwest Finland, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sjoros T, Saraste M, Matilainen M, Nylund M, Koivumaki M, Kuhle J, Leppert D, Airas L. Serum glial fibrillary acid protein associates with TSPO-expressing lesions in multiple sclerosis brain. Ther Adv Neurol Disord. 2025 Jul 28;18:17562864251352998. doi: 10.1177/17562864251352998. eCollection 2025. PMID 40756531